CLINICAL TRIAL: NCT00224926
Title: The Natural Course of Trichophyton Tonsurans Carriage and Infection: A Molecular and Biochemical Evaluation
Status: Completed | Type: Observational
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Other Study IDs: PPRU 10704
Record Dates: First submitted 2005-09-21; First posted 2005-09-23 (Estimated); Last update posted 2011-09-19 (Estimated); Status verified 2011-09

CONDITIONS: Tinea Capitis
Keywords: Tinea Capitis
MeSH Terms: conditions — Tinea Capitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — fungal scalp cultures
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Scalp Brushing — sterile, soft-head toothbrush massaged on scalp

SUMMARY:
To explore carrier and infection status of T.tonsurans tinea capitis and characterize the host-pathogen interaction as it relates to the disease presentation. The general hypothesis for this study is as follows: the type of genotypic and phenotypic variant to which a child is exposed accounts for the presentation status observed in Trichophyton tonsurans infection.The global outcome of this investigation is to reveal potential new drug targets designed to improve treatment outcomes in these children.

DETAILED DESCRIPTION:
Tinea capitis is an overwhelmingly prevalent disease of childhood estimated to be present in approximately 1 in 20 children at any point in time with an equal number of children serving as carriers of the fungal pathogen. Despite the widespread nature of the disease, the natural course of the infection remains incompletely described. The study will be driven by the following hypothesis: the type of genotypic and phenotypic variant to which a child is exposed accounts for the presentation status observed in Trichophyton tonsurans infection.

A fungal scalp culture will be acquired from all participants using a brush culture technique. Samples will be collected once a month over a two year time period.

ELIGIBILITY:
Inclusion Criteria:

* Preschool aged children will be eligible.

Exclusion Criteria:

* None

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: preschool aged children
Sampling Method: Probability Sample
Enrollment: 446 (Actual)
Dates: Start 2003-09; Study Completion 2005-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Rahman, PharmD, Principal Investigator — Children's Mercy Hosptials and Clinics
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States